CLINICAL TRIAL: NCT05551598
Title: A Randomized, Double-blind, Placebo-controlled Phase Ⅱ Clinical Study to Evaluate the Efficacy and Safety of Mitoxantrone Hydrochloride Liposome Injection in the Treatment of Neuromyelitis Optica Spectrum Disorder (NMOSD)
Brief Title: Efficacy and Safety of Mitoxantrone Hydrochloride Liposome Injection in the Treatment of Neuromyelitis Optica Spectrum Disorder (NMOSD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HE071-CSP-028
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2022-07

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mitoxantrone Hydrochloride Liposome Injection 8 mg/m^2 group (Experimental)
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection
- Mitoxantrone Hydrochloride Liposome Injection 12 mg/m^2 group (Experimental)
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection
- Placebo Injection every 12 weeks (Q12W). (Placebo Comparator)
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome Injection — IV, once every 12 weeks (Q12W)

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase Ⅱ study to evaluate the efficacy and safety of Mitoxantrone Hydrochloride Liposome Injection with different doses in participants with neuromyelitis optica spectrum disorder (NMOSD). Participants will be randomly enrolled into three groups: Mitoxantrone Hydrochloride Liposome Injection 8 mg/m^2 group, Mitoxantrone Hydrochloride Liposome Injection 12 mg/m^2 group, and Placebo group. The primary outcome measure is time to first protocol-defined relapse.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years (inclusive) at the time of signing the informed consent form, both men and women;
2. Participants meet the 2015 international consensus diagnostic criteria for neuromyelitis optica spectrum disease (NMOSD) and are AQP4-IgG positive or negative (acceptable test results within 24 weeks before signing the informed consent form);
3. Experienced at least 2 attacks within 1 year before screening and/or at least 3 relapses in the past 24 months, but have at least 1 documented clinical evidence of attack or relapse (including the first attack) within 12 months before screening;
4. Expanded disability status scale (EDSS) ≤ 7.5 points at screening and baseline retest;
5. Participants voluntarily sign the informed consent form and voluntarily complete the trial according to the protocol requirements.

Exclusion Criteria:

1. Pregnant or lactating female participants, or participants planning to have a child during the study;
2. Any surgical procedure within 4 weeks before randomization, with evidence of other demyelinating diseases or progressive multifocal leukoencephalopathy (PML);
3. Known active infection (excluding nail bed fungal infection or dental caries) within 4 weeks before randomization;
4. Hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody, or human immunodeficiency virus (HIV antibody) is positive;
5. History of drug or alcohol abuse or mental disorder within 1 year before randomization;
6. Evidence of active tuberculosis (TB; excluding patients receiving drugs to prevent latent TB infection);
7. Evidence of active interstitial lung disease;
8. Receipt of any live or live attenuated vaccine within 6 weeks before randomization;
9. History of malignancy, including solid tumors, hematological malignancies, and carcinoma in situ (except completely resected and cured basal cell carcinoma and squamous cell carcinoma or cervical carcinoma in situ) within the past 5 years;
10. History of severe drug allergy, allergy or intolerance to Mitoxantrone and liposomes (shock, allergic reactions);
11. Participants with other chronic active immune system diseases other than NMOSD or stable disease but requiring high-dose glucocorticoid maintenance therapy: such as rheumatoid arthritis, scleroderma, Schogren' s syndrome, ulcerative colitis, genetic immunodeficiency or drug-induced immunodeficiency; participants with positive autoantibodies only but without clinical manifestations can be enrolled in the trial;
12. Participants with other diseases not suitable for this study as judged by the investigator;
13. Received any investigational agent within 3 months prior to randomization, or participated in a medical device clinical study and judged by the investigator to have a potential impact on the results of this trial;
14. History of prior NMOSD therapy with any of the following: a. received prior mitoxantrone or anthracycline therapy, total body irradiation, or bone marrow transplantation at any time; b. received rituximab or any experimental B-cell depleting agent within 6 months prior to randomization, unless the participant had a B-cell count higher than LLN in the central laboratory; c. used any of the following within 3 months prior to randomization: Satralizumab,Tocilizumab,inebilizumab,Eculizumab,Alemtuzumab,Ciclosporin,Azathioprine,Cyclophosphamide,Tacrolimus,Mycophenolate mofetil. Any other treatment to prevent relapses in multiple sclerosis (MS) (eg, Interferon, Natalizumab, Glatiramer acetate, Fingolimod, Teriflunomide, or Dimethyl fumarate); d. intravenous immunoglobulin (IVIG) therapy, plasma exchange therapy (PE) within 1 month prior to randomization; e. participants who are receiving oral corticosteroids at doses higher than 30 mg/day in prednisolone conversion; f. anti-CD4, cladribine within 2 years prior to randomization.
15. Presence of the following clinically significant diseases: a. cardiac ejection fraction (EF) less than 50% by echocardiography or lower than the lower limit of laboratory values at the study site; history of chronic congestive heart failure, cardiac function NYHA class Ш ~ Ⅳ; b. any of the following events within 3 months before randomization: myocardial infarction, acute coronary syndrome, viral myocarditis, pulmonary embolism, stroke; coronary revascularization within 6 months; c. screening ECG showed QTc interval > 480 ms (according to Fridericia correction formula, QTc = QT/RR^0.33), or a history of severe QTc prolongation.
16. Patients with the following abnormalities in laboratory values during screening: a. aspartate aminotransferase (AST) > 3 × upper limit of normal (ULN), alanine aminotransferase (ALT) > 3 × ULN, total bilirubin > 1.5 × ULN (unless due to Gilbert 's syndrome); b. platelet count < 50,000/μL (or < 50 × 10^9/L), hemoglobin < 9 g/dL (or < 90 g/L), white blood cells < 2.0 × 10^3/μL, absolute neutrophil count < 1.0 × 10^3/μL; c. creatinine clearance (CLcr) < 60 mL/min (calculated using the Cockcroft-Gault formula: [140 - age (years)] × [body weight (kg)] × (0.85, if female)/[72 × serum creatinine (mg/dL)]) or receiving dialysis during screening;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Time to First Protocol-defined Relapse | Up to Week 48
  Time to First Protocol-defined Relapse was defined as time from randomization to first occurrence of relapse. Protocol-defined relapse was occurrence of new or worsening neurological symptoms attributable to neuromyelitis optica spectrum disorder (NMOSD).

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No